CLINICAL TRIAL: NCT06827652
Title: Observational Prospective Study of Individuals with Abdominal Aortic Aneurysm (AAA) to Monitor AAA Growth and Rupture Risk.
Brief Title: Triple-A Barcelona Study
Acronym: TABS
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-OMI-2019-102
Record Dates: First submitted 2025-01-23; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aneurysm, Aorta, risk
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted DNA and RNA extracted from blood cells, along with plasma samples will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Triple-A Barcelona Study (TABS), is a new hospital-based longitudinal study recruiting consecutive individuals with Abdominal Aortic Aneurysm (AAA) in Barcelona. Individuals that have at least one measurement of the abdominal aortic diameter, either by computed tomography scan or by ultrasound, along with anthropometric, clinical information, and blood samples for most follow-up visits are recruited.

DETAILED DESCRIPTION:
The Triple-A Barcelona Study (TABS) is a prospective longitudinal registry started in 2019. All individuals identified incidentally with AAA, defined as those with dilation in infrarenal abdominal aorta with a diameter greater than 30 mm13 that visit the Vascular and Endovascular Surgery Units of Hospital de la Santa Creu i Sant Pau and Hospital del Mar (Barcelona, Spain) from 2020 to the present are invited to participate to the project. Patients who did not consent to participation were not considered for enrollment. Upon enrollment, participant's medical history was carefully reviewed, and all previous measures of aortic diameter and available clinical information was included retrospectively in the database. All participants have at least one measurement of the abdominal aortic diameter, either by computed tomography scan (CT-scan) or by ultrasound along with anthropometric and clinical information, and blood samples for most follow-up visits. The first measurement was considered as the baseline. All measurements following the baseline measurement were used until aortic repair or rupture, or death. Individuals that were excluded from surgery after they exceeded the surgical threshold (due to concomitant pathology, AAA anatomy or patient rejection to surgery) were also considered for inclusion, and their retrospective data, if existing, was recorded. All patients were asked for an informed consent to participate in this study, and to be included in a clinical database. Type B dissections that progress to AAA, saccular aneurysms, mycotic aneurysms, visceral aneurysms or thoracic aneurysms were excluded. Aortic diameter was assessed using either ultrasound or CT-scan images.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of abdominal aortic aneurysm
* infrarenal abdominal aortic diameter greater than 30 mm

Exclusion Criteria:

* Type B dissections that progress to AAA
* saccular aneurysms
* mycotic aneurysms
* visceral aneurysms
* thoracic aneurysms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Individuals with a diagnosis of AAA visiting at Hospital de Sant Pau or Hospital del Mar in Barcelona.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal Aortic diameter | baseline, through study completion (every 2 years on average), pre-surgery
  Diameter in mm

CONTACTS AND LOCATIONS:
Overall Officials: Maria Sabater-Lleal, PhD, Principal Investigator — RESEARCH INSTITUTE/HOSP/SANTA CREU/PAU
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No